CLINICAL TRIAL: NCT00602186
Title: Effect of Tamsulosin vs Prazosin in Treatment of Female Voiding Dysfunction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tabriz University (Other)
Responsible Party: Lily Nosraty, Tabriz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 85-1
Record Dates: First submitted 2007-04-18; First posted 2008-01-28 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Neurogenic Bladder
Keywords: female voiding dysfunction; Tamsolusin; prazosin
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — Tamsulosin; Prazosin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): taking Tamsulosin
  Interventions: Drug: tamsolusin
- 2 (Active Comparator): taking prasosin
  Interventions: Drug: prazosin

INTERVENTIONS:
Drug: tamsolusin — 0.4 mg /day
  Other Names: Flomax
  Arms: 1
Drug: prazosin — 1 mg/day
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Tamsolusin or Prazosin are effective in the treatment of female voiding dysfunction(BOO)

DETAILED DESCRIPTION:
Voiding dysfunction is not uncommon in Tabriz.About 20% of patients in female urology clinic of Tabriz university of medical sciences sufered from some degrees of voiding dysfunction (due to bladder imparement or bladder outlet obstruction).There is limited information about medical treatment of those patients. On the other hand alpha adrenergic blockers are the first choice medication in BENIGN PROSTATIC HYPERPLASIA. There is some new facts about destribution of alpha adrenergic blockers in female pelvic floor.The purpose of this study is to comparision whether Tamsolusin 0.4/daily or Prazosin 1 mg/daily are effective in the treatment of female voiding dysfunction(BOO)

ELIGIBILITY:
Inclusion Criteria:

* Healthy females with voiding difficulty with MFR<12 and post void residual urine>50cc

Exclusion Criteria:

* History of pelvic floor surgury during last 3 month
* Any contraindication for Tamsolusin or prazosin

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-07; Primary Completion 2007-03 (Estimated); Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
patient symptoms improvement(Standard questionare) | every month untile 3 months

SECONDARY OUTCOMES:
Urodynamics parameters improvement | three months later

CONTACTS AND LOCATIONS:
Overall Officials: SAKINEH hajebrahimi, MD, Study Director — Urology department ofTabriz University of Medical Sciences